CLINICAL TRIAL: NCT01432197
Title: Occupational Therapy for Cancer Patients: A Randomised Controlled Study
Brief Title: Occupational Therapy for Cancer Patients: a Randomised, Controlled Study
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: University of Southern Denmark (Other)
Collaborators: Naestved Hospital (Other)
Responsible Party: Principal Investigator, Line Lindahl, Ph.D student, OT, MPH, University of Southern Denmark
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: RCT Occup Cancer
Record Dates: First submitted 2011-09-08; First posted 2011-09-12 (Estimated); Last update posted 2011-09-12 (Estimated); Status verified 2011-09

CONDITIONS: HRQOL (Health Related Quality of Life)
Keywords: HRQOL; Occupational therapy; ADL intervention; Cancer patients

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Occupational therapy intervention (Experimental): Intervention group: Standard treatment and care added with an ADL intervention program: 1) ADL training, 2) home modifications, 3) delivery and supervision in adaptive equipments, and 4) instruction in self-training programs.
  Control group: Standard treatment and care. No occupational therapy intervention.
  Interventions: Other: ADL intervention
- Standard treatment and care (No Intervention): Control group: Standard treatment and care. No occupational therapy intervention.

INTERVENTIONS:
Other: ADL intervention — 1) ADL training, 2) home modifications, 3) delivery and supervision in adaptive equipments, and 4) instruction in self-training programs.
  Arms: Occupational therapy intervention

SUMMARY:
The aim of this study is to investigate the effect of occupational therapy, in shape of activities of daily living, for cancer patients.

DETAILED DESCRIPTION:
Background

Cancer patients often experience serious dysfunctions leading to problems with activities of daily living (ADL) and reduced quality of life. Occupational therapy is believed to be effective in handling many of the problems with ADL experienced by patients with cancer, but the evidence is sparse.

Aim

The purpose of this study is to analyse the effects of an occupational therapy intervention targeting cancer patients.

Outcome measures are the patients self-reported quality of life and the patients ability to perform ADL.

Methods

Randomised controlled trial with 288 patients with cancer treated at Naestved hospital in Denmark. Occupational therapy intervention programme for the intervention group (N=144) and standard treatment and care for the controls (N=144).

A systematic review including studies of ADL intervention for cancer patients will be carried out. Feasibility of the recruitment and the intervention will be analysed and published.

The patients need for occupational therapy will be analysed using baseline information from the randomised controlled trial.

The effects of the intervention will be analysed using patient validated questionnaires including EORTC QLQ-C30 and the ADL taxonomy questionnaire.

ELIGIBILITY:
Inclusion Criteria:

* Cancer patients
* Disability comparable with a performance status of 10 to 70 on Karnofsky Performance Status Scale
* Able to read and understand Danish

Exclusion Criteria:

* Referred to occupational therapy before study start

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 116 (Actual)
Dates: Start 2010-03; Primary Completion 2011-06 (Actual)

PRIMARY OUTCOMES:
Health related quality of life | 15 months

SECONDARY OUTCOMES:
Ability to perform activities of daily living | 15 months

CONTACTS AND LOCATIONS:
Overall Officials: Dorte Gilsaa Hansen, Ph.D, M.D., Principal Investigator — Research Unit of General Practice, IST, University of Southern Denmark; Karen la Cour, Ph.D, OT, MSc, Principal Investigator — Health, Man and Society, IST, University of Southern Denmark
Locations (1):
- Research Unit of General Practice, IST, University of Southern Denmark, Odense, Denmark